CLINICAL TRIAL: NCT01850615
Title: Efficacy and Safety of FIAsp in a Basal-bolus Regimen Versus Basal Insulin Therapy, Both in Combination With Metformin in Adult Subjects With Type 2 Diabetes
Acronym: onset® 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1218-4049; 2012-005583-10 (EudraCT Number); U1111-1137-6242 (Other: WHO); CTRI/2014/01/004289 (Registry Identifier: Clinical Trials Registry - India (CTRI))
Record Dates: First submitted 2013-04-17; First posted 2013-05-09 (Estimated); Results first posted 2018-01-17 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FIAsp and basal insulin + metformin (Experimental): Subjects will receive FIAsp combined with their pre-trial basal insulin (insulin human, insulin detemir or insulin glargine) treatment in combination with their pre-trial metformin.
  Interventions: Drug: Faster-acting insulin aspart; Drug: basal insulin
- Basal insulin + metformin (Active Comparator): Subjects will continue their pre-trial basal insulin (insulin human, insulin detemir or insulin glargine) treatment in combination with their pre-trial metformin.
  Interventions: Drug: basal insulin

INTERVENTIONS:
Drug: Faster-acting insulin aspart — Administrated subcutaneously (s.c., under the skin) at each main meal.
  Other Names: NN1218
  Arms: FIAsp and basal insulin + metformin
Drug: basal insulin — Administrated subcutaneously (s.c., under the skin) once daily.

SUMMARY:
This trial is conducted in Asia, Europe, South America, and the United States of America (USA).

The aim of the trial is to investigate efficacy and safety of FIAsp in a basal-bolus regimen versus basal insulin therapy, both in combination with metformin in adult subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (diagnosed clinically) for at least 6 months prior to the screening visit (Visit 1)
* Current treatment with once daily insulin detemir, insulin glargine or human isophane insulin, NPH for at least 3 months prior to the screening visit (Visit 1)
* Current treatment with a) metformin with unchanged dosing for at least 3 months prior to screening (visit 1). The metformin dose must be at least 1000 mg or b) metformin in combination with sulfonylurea (SU) or glinide or Dipeptidyl peptidase-IV inhibitors and/or alpha-glucosidase inhibitors (AGI) with unchanged dosing for at least 3 months prior to screening (visit 1). The metformin dose must be at least 1000 mg
* HbA1c by central laboratory a) 7.5-9.5% (58 - 80 mmol/mol) (both inclusive) in the metformin group at the screening visit (Visit 1) or b) 7.5-9.0% (58 - 75 mmol/mol) (both inclusive) in the metformin + other oral antidiabetic drug (OAD) (sulphonylurea (SU), glinide, dipeptidyl peptidase-IV (DDP-IV) inhibitors, alpha-glucosidase inhibitors (AGI) combination group at the screening visit (Visit 1)
* Body mass index (BMI) equal or less than 40.0 kg/m^2

Exclusion Criteria:

* Any use of bolus insulin, except short-term use due to intermittent illness (no longer than 14 days of consecutive treatment) and not within 3 months prior to the screening visit (Visit 1)
* Use of Glucagon-like peptide-1 (GLP-1) agonists and/or Thiazolidinediones (TZD) within the last 3 months prior to screening (visit 1)
* Recurrent severe hypoglycaemia (more than one severe hypoglycaemic event during the last 12 months) or hypoglycaemic unawareness as judged by the Investigator, or hospitalisation for diabetic ketoacidosis during the previous 6 months prior to screening (Visit 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2013-09-23 (Actual); Primary Completion 2014-11-17 (Actual); Study Completion 2014-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (53):
- United States (30):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Peoria, Arizona
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, Santa Ana, California
  - Novo Nordisk Investigational Site, Tarzana, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Conyers, Georgia
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Kalamazoo, Michigan
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Henderson, Nevada
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Brooklyn, New York
  - Novo Nordisk Investigational Site, Asheboro, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Downingtown, Pennsylvania
  - Novo Nordisk Investigational Site, Reading, Pennsylvania
  - Novo Nordisk Investigational Site, Greenville, South Carolina
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Ogden, Utah
- Argentina (5):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Capital Federal
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Godoy Cruz
  - Novo Nordisk Investigational Site, San Isidro
- India (7):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Visakhapatnam, Andhra Pradesh
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Chandigarh, Punjab
  - Novo Nordisk Investigational Site, Coimbatore, Tamil Nadu
- Mexico (2):
  - Novo Nordisk Investigational Site, Guadalajara, Jalisco
  - Novo Nordisk Investigational Site, Mexico City, México, D.F.
- Romania (5):
  - Novo Nordisk Investigational Site, Târgu Mureş, Mureș County
  - Novo Nordisk Investigational Site, Ploieşti, Prahova
  - Novo Nordisk Investigational Site, Timișoara, Timiș County
  - Novo Nordisk Investigational Site, Brasov
  - Novo Nordisk Investigational Site, Suceava
- Slovenia (4):
  - Novo Nordisk Investigational Site, Brežice
  - Novo Nordisk Investigational Site, Koper
  - Novo Nordisk Investigational Site, Kranj
  - Novo Nordisk Investigational Site, Novo Mesto

REFERENCES:
- [Background] Peters AL, Piletic M, Ejstrud J, Salvesen-Sykes K, Snyder J, Bowering K. Baseline nocturnal glucose change: A predictor of the treatment effect of bolus intensification in insulin-treated type 2 diabetes. Diabetes Obes Metab. 2019 Jul;21(7):1752-1756. doi: 10.1111/dom.13729. Epub 2019 Apr 23. PMID 30924578
- [Result] Rodbard HW, Tripathy D, Vidrio Velazquez M, Demissie M, Tamer SC, Piletic M. Adding fast-acting insulin aspart to basal insulin significantly improved glycaemic control in patients with type 2 diabetes: A randomized, 18-week, open-label, phase 3 trial (onset 3). Diabetes Obes Metab. 2017 Oct;19(10):1389-1396. doi: 10.1111/dom.12955. Epub 2017 Jul 6. PMID 28345792
- [Result] Heller S, Bowering K, Raskin P, Liebl A, Buchholtz K, Gorst-Rasmussen A, Pieber TR. The effect of basal-bolus therapy varies with baseline 1,5-anhydroglucitol level in people with Type 2 diabetes: a post hoc analysis. Diabet Med. 2018 May 26;35(9):1273-8. doi: 10.1111/dme.13693. Online ahead of print. PMID 29802636
- [Result] Bowering K, Rodbard HW, Russell-Jones D, Bode B, Harris S, Piletic M, Heller S, Woo V, Babu V, Dethlefsen C, Mathieu C. Investigating the Association Between Baseline Characteristics (HbA1c and Body Mass Index) and Clinical Outcomes of Fast-Acting Insulin Aspart in People with Diabetes: A Post Hoc Analysis. Diabetes Ther. 2019 Feb;10(1):177-188. doi: 10.1007/s13300-018-0553-7. Epub 2018 Dec 13. PMID 30547388
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 51 sites in 6 countries as follows: Argentina: 4 sites; India: 8 sites; Mexico: 3 sites; Romania: 5 sites; Slovenia: 4 sites; United States: 27 sites.
Pre-assignment Details: A total of 555 subjects were screened, of which 232 subjects were screening failures and 323 subjects were enrolled and entered the run-in (pre-assignment) period. Of those, 87 subjects were run-in failures. Hence, 236 subjects were randomized to the 18 weeks of treatment period.
Groups:
- Faster Aspart + Basal: During the 18-week treatment period, subjects received subcutaneous (s.c., under the skin) injection of faster aspart (bolus insulin) along with s.c. basal insulin (insulin detemir or insulin glargine or NPH insulin) and metformin. Treatment recommendations were developed for the different trial products specifying the recommended dose adjustments at different plasma glucose (PG) levels. Trial products were titrated according to the insulin dosing recommendations provided during the study. No maximum dose of insulin was specified as doses were titrated individually. Faster aspart was administered 0-2 minutes before each main meal (i.e., breakfast, lunch and main evening meal). The basal insulin injection was to be given once daily (OD), in the evening, at approximately the same time each day.
- Basal: During the 18-week treatment period, subjects received s.c. injection of basal insulin (insulin detemir or insulin glargine or NPH insulin) and metformin. Treatment recommendations were developed for the different trial products specifying the recommended dose adjustments at different PG levels. Trial products were titrated according to the insulin dosing recommendations provided during the study. No maximum dose of insulin was specified as doses were titrated individually. The basal insulin injection was to be given OD, in the evening, at approximately the same time each day.
Period: Overall Study
Arm/Group | Faster Aspart + Basal | Basal
Started | 116 | 120
Exposed | 115 | 120
Completed | 107 | 115
Not Completed | 9 | 5
Not completed — Protocol Violation | 4 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Unclassified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised subjects
Groups:
- Faster Aspart + Basal: During the 18-week treatment period, subjects received subcutaneous (s.c., under the skin) injection of faster aspart (bolus insulin) along with s.c. basal insulin (insulin detemir or insulin glargine or NPH insulin) and metformin. Treatment recommendations were developed for the different trial products specifying the recommended dose adjustments at different PG levels. Trial products were titrated according to the insulin dosing recommendations provided during the study. No maximum dose of insulin was specified as doses were titrated individually. Faster aspart was administered 0-2 minutes before each main meal (i.e., breakfast, lunch and main evening meal). The basal insulin injection was to be given OD, in the evening, at approximately the same time each day.
- Basal: During the 18-week treatment period, subjects received s.c. injection of basal insulin (insulin detemir or insulin glargine or NPH insulin) and metformin. Treatment recommendations were developed for the different trial products specifying the recommended dose adjustments at different (PG) levels. Trial products were titrated according to the insulin dosing recommendations provided during the study. No maximum dose of insulin was specified as doses were titrated individually. The basal insulin injection was to be given OD, in the evening, at approximately the same time each day.
- Total: Total of all reporting groups
Arm/Group | Faster Aspart + Basal | Basal | Total
Number analyzed (Participants) | 116 | 120 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (9.9) | 57.4 (8.5) | 57.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 61 | 122
  Male | 55 | 59 | 114
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin] | 7.93 (0.69) | 7.92 (0.68) | 7.93 (0.69)
Body weight [Mean (Standard Deviation); unit: Kg] | 82.2 (16.2) | 85.1 (17.3) | 83.7 (16.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c
Description: For this endpoint, baseline (week 0) and week 18 data are presented, where week 18 data are the "end of trial" data containing last available measurements.
Time Frame: Week 0, week 18
Population: Full analysis set included all randomised subjects.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin
Arm/Group | Faster Aspart + Basal | Basal
Number analyzed (Participants) | 116 | 120
Percentage of glycosylated haemoglobin
  Baseline | 7.93 (0.69) | 7.92 (0.68)
  Week 18 | 6.78 (0.92) | 7.7 (0.93)
Statistical Analysis 1: Comparison: Faster Aspart + Basal vs Basal; Change from baseline in HbA1c after 18 weeks of treatment was analysed using a mixed-effect model for repeated measurements (MMRM) where all calculated changes in HbA1c from baseline at visits 16, 22 and 28 were included in the analysis. This model included treatment, region and strata as fixed factors, subject as random effect, baseline HbA1c as covariate and interaction between all fixed effects and visit, and between the covariate and visit; Test type: Superiority or Other; Treatment difference = -0.94, 95% CI 2-sided [-1.17 to -0.72] — Superiority was considered confirmed if the upper bound of the two-sided 95% confidence interval (CI) for the estimated treatment difference (faster aspart+basal minus basal only), which was calculated using the FAS, was below 0%

2. Secondary Outcome: Self-measured Plasma Glucose (SMPG) 7-point Profile: Post Prandial Plasma Glucose (PPG), Overall 2-hour Mean (of Breakfast, Lunch, Main Evening Meal)
Description: For this endpoint the "end of trial" data containing last available measurements are presented. PPG measurements were recorded by the subjects at 2 hours after each meal (breakfast, lunch and main evening meal) as part of three 7-point profiles (SMPG) prior to the visits. Individual mean meal PPG (post-breakfast, post-lunch, post-main evening meal) was derived from the three measurements.
Time Frame: After 18 weeks of randomised treatment
Population: FAS included all randomised subjects. Number analysed for individual time-points = treatment wise number of subjects who contributed to analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart + Basal | Basal
Number analyzed (Participants) | 116 | 120
mmol/L
  PPG breakfast; SMPG: number analyzed (Participants) | 114 | 120
  PPG breakfast; SMPG | 7.2 (1.8) | 9 (2.4)
  PPG lunch; SMPG: number analyzed (Participants) | 114 | 120
  PPG lunch; SMPG | 7.1 (1.9) | 9.7 (2.6)
  PPG main evening meal; SMPG | 7.4 (1.9) | 10.1 (2.9)

3. Secondary Outcome: Self-measured Plasma Glucose (SMPG) 7-point Profile: Prandial Plasma Glucose (PG) Increment, Overall 2-hour Mean (of Breakfast, Lunch, Main Evening Meal)
Description: For this endpoint the "end of trial" data containing last available measurements are presented. Prandial PG increment for each meal (breakfast, lunch, main evening meal) was derived from the 7-point profiles (SMPG) as the difference between the PPG value 2 hours after each meal and the PG value before each meal. Individual mean meal PPG (post-breakfast, post-lunch, post-main evening meal) was derived from the three measurements.
Time Frame: After 18 weeks of randomised treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart + Basal | Basal
Number analyzed (Participants) | 116 | 120
mmol/L
  Breakfast increment; SMPG: number analyzed (Participants) | 114 | 120
  Breakfast increment; SMPG | 1.2 (1.8) | 2.9 (2.4)
  Lunch increment; SMPG: number analyzed (Participants) | 114 | 120
  Lunch increment; SMPG | 0.9 (2.0) | 1.8 (2.2)
  Main evening meal increment; SMPG: number analyzed (Participants) | 115 | 120
  Main evening meal increment; SMPG | 0.7 (1.7) | 1.4 (1.9)

4. Secondary Outcome: Change From Baseline in Body Weight
Description: as for outcome 1
Time Frame: Week 0, week 18
Population: FAS included all randomised subjects.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Faster Aspart + Basal | Basal
Number analyzed (Participants) | 116 | 120
Kg
  Baseline | 82.2 (16.2) | 85.1 (17.3)
  Week 18 | 83.9 (16.9) | 85.4 (17.5)

5. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes
Description: Plasma glucose (PG) was measured and recorded when a hypoglycaemic episode was suspected. All PG values ≤3.9 mmol/L (70 mg/dL) or >3.9 mmol/L (70 mg/dL) when they occurred in conjunction with hypoglycaemic symptoms were recorded by the subject. Numbers of treatment emergent hypoglycaemic episodes were recorded during 18 weeks of treatment.
Time Frame: Weeks 0-18
Population: The Safety Analysis Set (SAS) included all subjects receiving at least one dose of the investigational product or its comparator.
Measure: Number; unit: Number of episodes
Arm/Group | Faster Aspart + Basal | Basal
Number analyzed (Participants) | 115 | 120
Number of episodes | 1908 | 347

6. Secondary Outcome: Number of Adverse Events
Description: All adverse events (AEs) described here refer to treatment emergent adverse events (TEAE). A TEAE was defined as an event that had onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment, week 18.
Time Frame: Weeks 0-18
Population: The SAS included all subjects receiving at least one dose of the investigational product or its comparator.
Measure: Number; unit: Number of events
Arm/Group | Faster Aspart + Basal | Basal
Number analyzed (Participants) | 115 | 120
Number of events | 123 | 121

ADVERSE EVENTS:
Time Frame: During 18 weeks of randomised treatment period + 7 days of follow-up period.
Description: All AEs described here refer to TEAEs. The SAS included all subjects receiving at least one dose of the investigational product or its comparator.
Arm/Group | Faster Aspart + Basal | Basal
Serious Adverse Events (participants affected / at risk) | 6/115 | 5/120
Other Adverse Events (participants affected / at risk) | 2/115 | 6/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faster Aspart + Basal (N=115) | Basal (N=120)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Malignant respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wrong drug administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faster Aspart + Basal (N=115) | Basal (N=120)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.